CLINICAL TRIAL: NCT03394521
Title: Progression Evaluation in Glaucoma (PEG): Progression of Disease in Patients Newly Diagnosed With Glaucoma and Glaucoma Suspects Participating in the GATE Study
Brief Title: Progression of Disease in Patients Newly Diagnosed With Glaucoma and Glaucoma Suspects Participating in the GATE Study
Acronym: PEG
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Other Study IDs: 02/019/15
Record Dates: First submitted 2017-05-22; First posted 2018-01-09 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Glaucoma
Keywords: glaucoma suspect; ocular hypertension; progression
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Routine clinical practice — This is an observational study

SUMMARY:
The purpose of this study is to measure how many patients develop worsening glaucoma in the early years (2-4 years) of routine monitoring in hospital eye services. We will study a group of patients who were initially diagnosed as having glaucoma, or having high pressure in the eye (ocular hypertension) or having been diagnosed as a glaucoma suspect.

DETAILED DESCRIPTION:
In the UK, patients with possible signs of glaucoma or ocular hypertension (OHT) are usually picked up at a routine sight test at their optician or general practitioner. These patients are usually diagnosed in secondary care hospital eye services by an ophthalmologist.

In addition to those diagnosed with OHT and glaucoma there are a large group of patients who have ocular characteristics similar to those found in glaucoma patients, but could also represent variations in normality. In this group, 'glaucoma suspects', monitoring in secondary care for a number of years is recommended in order to establish whether they have glaucoma or if after several years of monitoring there are no clear signs of glaucoma the patient may be discharged.

In our study we will conduct a case-note review of a well-defined cohort of patients who were first identified through a diagnostic accuracy study (the GATE study). This includes (1) patients with OHT, (2) patients identified as glaucoma suspects and (3) patients diagnosed with glaucoma. We will investigate how many patients have experience worsening disease and how many patients have been discharged due to a low risk of glaucoma. We will also investigate the relationship between baseline demographic characteristics and characteristics of the eye and progression of disease.

ELIGIBILITY:
Eligibility for patients to be recruited into the GATE study was as follows:

Inclusion criteria:

- Adults referred from community optometrists or general practitioner to hospital eye services with suspected glaucoma, including those with ocular hypertension.

Exclusion criteria:

* Patients referred to hospital eye services because of other ocular disease;
* patients < 18 years old;
* patients who cannot give informed consent,
* patients already diagnosed with glaucoma.

This study cohort is further defined from the GATE population as

Selection criteria:

* GATE study patients with a baseline diagnosis of OHT, Glaucoma suspect or Glaucoma (any mechanism);
* remaining in secondary care monitoring after first visit;
* recruited at Aberdeen Royal Infirmary or Hinchingbrooke Hospital NHS Trust.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients identified through the GATE study - newly referred from community to hospital eye services with suspected glaucoma
Sampling Method: Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Development of glaucoma | 4 years
  Proportion of glaucoma suspects and OHT patients who develop glaucoma annually up to 4 years after diagnosis in secondary care

SECONDARY OUTCOMES:
Progression of glaucoma | 1,2,3,4 years
  Proportion of the cohort of glaucoma patients with progression of disease up to 4 years
Predictors of disease progression | 4 years
  Evaluation of predictors of disease progression from baseline demographic and ocular characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Katie Banister, Principal Investigator — University of Aberdeen

IPD SHARING:
Plan to Share IPD: Undecided